CLINICAL TRIAL: NCT04039217
Title: ART Persistence: Antiretroviral Drug Persistence in Different Body Compartments in HIV Negative Men Who Have Sex With Men
Brief Title: Antiretroviral Therapy (ART) Persistence in Different Body Compartments in HIV Negative MSM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Colleen Kelley, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00111410
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Results first posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-01

CONDITIONS: ART; HIV
Keywords: PrEP; PEP; MSM; Short-course regimen; Pharmacokinetics
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sample collection 2, 48, and 96 hours after first dose of Biktarvy (Experimental): Participants in this study arm (Arm A) will provide biological specimens 2, 48, and 96 hours after the in-clinic dose of Biktarvy. Approximately 24 mL of blood will be drawn, an oral cheek swab, 1 pre-wet penile swab and 1 dry penile swab, and a urethral swab will be collected. After previous swab collections are complete, participants will be asked to provide a urine sample (some of which will be used for gonorrhea and chlamydia testing). Participants will undergo rectal biopsy collection at one of the study visits.
  Interventions: Drug: Biktarvy
- Sample collection 4, 26, and 120 hours after first dose of Biktarvy (Experimental): Participants in this study arm (Arm B) will provide biological specimens 4, 26, and 120 hours after the in-clinic dose of Biktarvy. Approximately 24 mL of blood will be drawn, an oral cheek swab, 1 pre-wet penile swab and 1 dry penile swab, and a urethral swab will be collected. After previous swab collections are complete, participants will be asked to provide a urine sample (some of which will be used for gonorrhea and chlamydia testing). Participants will undergo rectal biopsy collection at one of the study visits.
  Interventions: Drug: Biktarvy
- Sample collection 24, 28, and 72 hours after first dose of Biktarvy (Experimental): Participants in this study arm (Arm C) will provide biological specimens 24, 28, and 72 hours after the in-clinic dose of Biktarvy. Approximately 24 mL of blood will be drawn, an oral cheek swab, 1 pre-wet penile swab and 1 dry penile swab, and a urethral swab will be collected. After previous swab collections are complete, participants will be asked to provide a urine sample (some of which will be used for gonorrhea and chlamydia testing). Participants will undergo rectal biopsy collection at one of the study visits.
  Interventions: Drug: Biktarvy

INTERVENTIONS:
Drug: Biktarvy — Participants will be given two doses of the oral fixed dose combination anti-HIV medication Biktarvy (BIC/FTC/TAF) separated by 24 hours. The first dose is given in the clinic and participants are instructed to take the second dose at home, 24 hours after the first dose.
  Other Names: BIC/FTC/TAF

SUMMARY:
The study seeks to understand how anti-HIV drug Biktarvy, which contains the drugs tenofovir alafenamide (TAF), emtricitabine (FTC), and bictegravir (BIC) is absorbed and how long it persists in different body compartments, including mucosal tissues, as it may be considered for PrEP or PEP regimens in the future.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) continue to be disproportionately affected by HIV. The majority of MSM acquire HIV after exposure to the rectal mucosa through receptive anal intercourse without condoms. Pre-exposure prophylaxis (PrEP) and post-exposure prophylaxis (PEP) are recommended for MSM who may be exposed to HIV to prevent infection. Current recommendations for PrEP are to take the combination anti-HIV drug, tenofovir+emtricitabine (TDF/FTC), on a daily basis for the duration of someone's HIV risk exposure period, which could be months or years. For PEP, a three-drug anti-HIV medication is recommended within 72 hours of a possible exposure for a 28-day course. While PrEP and PEP are effective, some people find it difficult to follow the recommended regimen. Therefore, additional short-course dosing regimens for PrEP and PEP are being considered for future development. The study drug provided in this study will not protect participants from HIV or treat any active infection. This proposal seeks to understand how other anti-HIV medications are absorbed and how long they persist in different body compartments, including mucosal tissues, as they may be considered for PrEP or PEP regimens in the future.

Participants will be sequentially enrolled into study arms. All participants will take two doses of Biktarvy and then will have biological samples collected at different time points. Blood will be collected at three different time points and a rectal biopsy will occur once. Participants may participate in more than one study arm or subgroup; however, at least 6 weeks must lapse after completion of one study arm or subgroup, before entry into another.

Median drug levels of TAF, FTC, and BIC in plasma, peripheral blood mononuclear cells (PBMCs) and rectal tissues will be calculated at baseline, 24 hours after the first dose and 120 hours after the first dose as the primary outcomes of this study. Samples collected at other time points will be stored for future exploratory analyses.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-negative man who reports receptive anal sex with another man in the last 6 months
2. Aged 18-49 years
3. Not currently taking PrEP and no plans to initiate during study
4. Not currently taking PEP
5. Able to provide informed consent in English
6. No plans for relocation in the next 3 months
7. Willing to undergo peripheral blood, penile swabs, urine, and rectal biopsy sampling
8. Willing to use study products as directed
9. Willing to abstain from receptive anal intercourse 3 days prior to starting study product and for the duration of the study and for 7 days after any rectal biopsy procedure.
10. Hepatitis B surface antigen (HBsAg) must be negative (screening lab test)
11. Creatine clearance >60 ml/min

Exclusion Criteria:

1. History of inflammatory bowel disease or other inflammatory, infiltrative, infectious or vascular condition involving the lower gastrointestinal tract that, in the judgment of the investigators, may be worsened by study procedures or may significantly distort the anatomy of the distal large bowel
2. Currently infected with hepatitis virus and/ or have liver disease
3. Current or chronic history of kidney disease
4. Significant laboratory abnormalities at baseline visit, including but not limited to:

   1. Hgb ≤ 10 g/dL
   2. partial thromboplastin time (PTT) > 1.5x upper limit of normal (ULN) or international normalized ratio (INR) > 1.5x ULN
   3. Platelet count <100,000
   4. Creatinine clearance <60
   5. HBsAg reactive
5. Any known medical condition that, in the judgment of the investigators, increases the risk of local or systemic complications of endoscopic procedures or pelvic examination, including but not limited to:

   1. Uncontrolled or severe cardiac arrhythmia
   2. Recent major abdominal, cardiothoracic, or neurological surgery
   3. History of uncontrolled bleeding diathesis
   4. History of colonic, rectal, fistula, or malignancy
   5. History or evidence on clinical examination of ulcerative, suppurative, or proliferative lesions of the anorectal mucosa, or untreated sexually transmitted disease with mucosal involvement
6. Continued need for, or use during the 14 days prior to enrollment, of the following medications:

   1. Aspirin or more than 4 doses of NSAIDs
   2. Warfarin, heparin (low-molecular weight or unfractionated), platelet aggregation inhibitors, or fibrinolytic agents
   3. Any form of rectally administered agent besides lubricants or douching used for sexual intercourse
7. Continued need for, or use during the 90 days prior to enrollment, of the following medications:

   1. Systemic immunomodulatory agents
   2. Supraphysiologic doses of steroids (short course steroids less than 7 days duration, allowable at the discretion of the investigators)
   3. Experimental medications, vaccines, or biologicals
8. Intent to use HIV antiretroviral pre/post-exposure prophylaxis (PrEP or PEP) during the study, outside of the study procedures
9. Symptoms of an untreated rectal sexually transmitted infection (e.g. rectal pain, discharge, bleeding, etc.)
10. Current use of hormonal therapy
11. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.
12. Participants taking potent inhibitors (e.g. itraconazole, diltiazem) or inducers (e.g. rifampin, phenytoin) of the CYP3A4 enzyme will be excluded from the study.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelley, MD, Principal Investigator — Emory University
Locations (1):
- Hope Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (e.g., text, tables, figures, and appendices), will be available for sharing.
Supporting Information: Study Protocol
Time Frame: Data will become available Beginning 9 months and ending at 36 months following publication to researchers who provide a methodologically sound proposal.
Access Criteria: Proposals should be directed to colleen.kelley@emory.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began on September 30, 2019 and all follow-up with participants was complete by August 28, 2020. Participants were enrolled at the Hope Clinic in Atlanta, Georgia, USA.
Pre-assignment Details: Enrollment began sequentially in Arm A, followed by Arms B and C. Arms A, B, and C were further broken down into two different sub-groups, determining the timing of the rectal biopsy procedure. Enrollment ended prior to enrolling Arm C.2. Participants were able to take part in multiple study arms, with at least 6 weeks after completion of one study arm before beginning another one. In total, 20 participants enrolled. Two individuals participated three times and one individual participated twice.
Groups:
- Biktarvy: Participants were given 2 doses of the oral fixed dose combination anti-HIV medication Biktarvy (BIC/FTC/TAF) separated by 24 hours, and had specimens collected at different time points.
  * Arm A.1: blood collection occurred 2, 48, and 96 hours after the in-clinic dose of Biktarvy; rectal biopsy occurred 2 hours after the in-clinic dose of Biktarvy
  * Arm A.2: blood collection occurred 2, 48, and 96 hours after the in-clinic dose of Biktarvy; rectal biopsy occurred 48 hours after the in-clinic dose of Biktarvy
  * Arm A.3: blood collection occurred 2, 48, and 96 hours after the in-clinic dose of Biktarvy; rectal biopsy occurred 96 hours after the in-clinic dose of Biktarvy
  * Arm B.1: blood collection occurred 4, 26, and 120 hours after the in-clinic dose of Biktarvy; rectal biopsy occurred 4 hours after the in-clinic dose of Biktarvy
  * Arm B.2: blood collection occurred 4, 26, and 120 hours after the in-clinic dose of Biktarvy; rectal biopsy occurred 120 hours after the in-clinic dose of Biktarvy
  * Arm C.1: blood collection occurred 24, 28, and 72 hours after the in-clinic dose of Biktarvy; rectal biopsy occurred 24 hours after the in-clinic dose of Biktarvy
  * Arm C.2: blood collection occurred 24, 28, and 72 hours after the in-clinic dose of Biktarvy; rectal biopsy occurred 72 hours after the in-clinic dose of Biktarvy
Period: Overall Study
Arm/Group | Biktarvy
Started | 20
Started Study Arm A.1 | 4
Completed Study Arm A.1 | 4
Started Study Arm A.2 | 4
Completed Study Arm A.2 | 4
Started Study Arm A.3 | 4
Completed Study Arm A.3 | 4
Started Study Arm B.1 | 4
Completed Study Arm B.1 | 4
Started Study Arm B.2 | 4
Completed Study Arm B.2 | 4
Started Study Arm C.1 | 5
Completed Study Arm C.1 | 4
Started Study Arm C.2 | 0
Completed Study Arm C.2 | 0
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Biktarvy: Participants were given two doses of the oral fixed dose combination anti-HIV medication Biktarvy (BIC/FTC/TAF) separated by 24 hours, and had specimens collected at different time points.
Arm/Group | Biktarvy
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.11 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Median Drug Levels in Plasma
Description: Median drug levels of tenofovir (TFV), emtricitabine (FTC), and bictegravir (BIC) in plasma were determined. Concentrations below the limit of quantification (LOQ) are assigned a value of zero. The prespecified outcomes of interest are plasma concentrations of the components of Biktarvy at 24 and 120 hours after the initial dose. All other time points of sample collection are for future exploratory analyses and have not been analyzed. Only the time points of sample collection that were prespecified as primary study outcomes are presented here.
Time Frame: Baseline (pre-dosing), 24 hours after the first dose, and 120 hours after first dose
Population: This analysis includes participants with usable samples at the indicated time points. Only the collection times of 24 and 120 hours post-dosing were prespecified for reporting.
Measure: Median (Full Range); unit: ng/mL
Groups:
- Sample Collection 2, 48, and 96 Hours After First Dose of Biktarvy: Participants in study Arm A provided biological specimens 2, 48, and 96 hours after the in-clinic dose of Biktarvy. Participants had a rectal biopsy at one of the study visits.
- Sample Collection 4, 26, and 120 Hours After First Dose of Biktarvy: Participants in study Arm B provided biological specimens 4, 26, and 120 hours after the in-clinic dose of Biktarvy. Participants also had a rectal biopsy at one of the study visits.
- Sample Collection 24, 28, and 72 Hours After First Dose of Biktarvy: Participants in study Arm C will provide biological specimens 24, 28, and 72 hours after the in-clinic dose of Biktarvy. Participants also had a rectal biopsy at one of the study visits.
Arm/Group | Sample Collection 2, 48, and 96 Hours After First Dose of Biktarvy | Sample Collection 4, 26, and 120 Hours After First Dose of Biktarvy | Sample Collection 24, 28, and 72 Hours After First Dose of Biktarvy
Number analyzed (Participants) | 4 | 4 | 4
ng/mL
  TFV at Baseline (pre-dosing) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  TFV at 24 hours after the first dose: number analyzed (Participants) | 0 | 0 | 4
  TFV at 24 hours after the first dose |  |  | 0 [0 to 0]
  TFV at 120 hours after first dose: number analyzed (Participants) | 0 | 4 | 0
  TFV at 120 hours after first dose |  | 0 [0 to 0] |
  FTC at Baseline (pre-dosing) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  FTC at 24 hours after the first dose: number analyzed (Participants) | 0 | 0 | 4
  FTC at 24 hours after the first dose |  |  | 33 [25 to 42]
  FTC at 120 hours after first dose: number analyzed (Participants) | 0 | 4 | 0
  FTC at 120 hours after first dose |  | 0 [0 to 0] |
  BIC at Baseline (pre-dosing) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  BIC at 24 hours after the first dose: number analyzed (Participants) | 0 | 0 | 4
  BIC at 24 hours after the first dose |  |  | 1296 [623 to 1698]
  BIC at 120 hours after first dose: number analyzed (Participants) | 0 | 4 | 0
  BIC at 120 hours after first dose |  | 267 [130 to 559] |

2. Primary Outcome: Median Drug Concentration in Peripheral Blood Mononuclear Cells (PBMCs)
Description: Median drug concentrations of tenofovir-diphosphate (TFV-DP) and emtricitabine-triphosphate (FTC-TP) in PBMCs were determined. Concentrations below the limit of quantification (LOQ) are assigned a value of zero. The prespecified outcomes of interest are PBMC concentrations of the components of Biktarvy at 24 and 120 hours after the initial dose. All other time points of sample collection are for future exploratory analyses and have not been analyzed. Only the time points of sample collection that were prespecified as primary study outcomes are presented here.
Time Frame: Baseline (pre-dosing), 24 hours after the first dose, and 120 hours after first dose
Population: This analysis includes participants with usable samples at the indicated time points. Only the collection times of 24 and 120 hours post-dosing were prespecified for reporting. Technical difficulties precluded the TFV-DP and FTC-TP measures in PBMCs for a large number of samples and therefore, data are not available for all drugs for all participants at these time points.
Measure: Median (Full Range); unit: fmol/10^6 cells
Arm/Group | Sample Collection 2, 48, and 96 Hours After First Dose of Biktarvy | Sample Collection 4, 26, and 120 Hours After First Dose of Biktarvy | Sample Collection 24, 28, and 72 Hours After First Dose of Biktarvy
Number analyzed (Participants) | 3 | 3 | 3
fmol/10^6 cells
  TFV-DP at Baseline (pre-dosing) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  TFV-DP at 24 hours after the first dose: number analyzed (Participants) | 0 | 0 | 3
  TFV-DP at 24 hours after the first dose |  |  | 98 [73 to 239]
  TFV-DP at 120 hours after first dose: number analyzed (Participants) | 0 | 3 | 0
  TFV-DP at 120 hours after first dose |  | 189 [136 to 273] |
  FTC-TP at Baseline (pre-dosing) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  FTC-TP at 24 hours after the first dose: number analyzed (Participants) | 0 | 0 | 3
  FTC-TP at 24 hours after the first dose |  |  | 3450 [1723 to 4910]
  FTC-TP at 120 hours after first dose: number analyzed (Participants) | 0 | 3 | 0
  FTC-TP at 120 hours after first dose |  | 1966 [1268 to 2168] |

3. Primary Outcome: Median Drug Levels in Rectal Tissues
Description: Median drug levels of TFV, FTC, and BIC in rectal tissue were determined. Concentrations below the limit of quantification (LOQ) are assigned a value of zero. The prespecified outcomes of interest are rectal tissue concentrations of the components of Biktarvy at 24 and 120 hours after the initial dose. All other time points of sample collection are for future exploratory analyses and have not been analyzed. Only the time points of sample collection that were prespecified as primary study outcomes are presented here.
Time Frame: Baseline (pre-dosing), 24 hours after the first dose, and 120 hours after first dose
Population: This analysis includes participants with usable samples at the indicated time points. Only the collection times of 24 and 120 hours post-dosing were prespecified for reporting. Technical difficulties precluded the drug measures in rectal tissues for a large number of samples and therefore, data are not available for all drugs for all participants at these time points.
Measure: Median (Full Range); unit: ng/mg
Arm/Group | Sample Collection 2, 48, and 96 Hours After First Dose of Biktarvy | Sample Collection 4, 26, and 120 Hours After First Dose of Biktarvy | Sample Collection 24, 28, and 72 Hours After First Dose of Biktarvy
Number analyzed (Participants) | 4 | 4 | 4
ng/mg
  TFV at Baseline (pre-dosing) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  TFV at 24 hours after the first dose: number analyzed (Participants) | 0 | 0 | 4
  TFV at 24 hours after the first dose |  |  | 0 [0 to 0.052]
  TFV at 120 hours after first dose: number analyzed (Participants) | 0 | 4 | 0
  TFV at 120 hours after first dose |  | 0 [0 to 0.052] |
  FTC at Baseline (pre-dosing) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  FTC at 24 hours after the first dose: number analyzed (Participants) | 0 | 0 | 4
  FTC at 24 hours after the first dose |  |  | 0.233 [0.025 to 0.440]
  FTC at 120 hours after first dose: number analyzed (Participants) | 0 | 4 | 0
  FTC at 120 hours after first dose |  | 0.064 [0 to 0.094] |
  BIC at Baseline (pre-dosing) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  BIC at 24 hours after the first dose: number analyzed (Participants) | 0 | 0 | 4
  BIC at 24 hours after the first dose |  |  | 0.105 [0.030 to 0.521]
  BIC at 120 hours after first dose: number analyzed (Participants) | 0 | 4 | 0
  BIC at 120 hours after first dose |  | 0.020 [0 to 0.035] |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the study visit where the first dose of medication was given through two days after the rectal biopsy was performed (up to 7 days).
Arm/Group | Sample Collection 2, 48, and 96 Hours After First Dose of Biktarvy | Sample Collection 4, 26, and 120 Hours After First Dose of Biktarvy | Sample Collection 24, 28, and 72 Hours After First Dose of Biktarvy
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT04039217/Prot_SAP_000.pdf